CLINICAL TRIAL: NCT01963949
Title: Prospective, Observational Study of Biomarkers in Liver Cancer - Identification of Actionable Events
Status: Withdrawn | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: SCCC
Record Dates: First submitted 2013-10-11; First posted 2013-10-17 (Estimated); Last update posted 2014-05-19 (Estimated); Status verified 2014-05

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples Without DNA — To collect tumor tissue from patients with liver masses suspicious for primary liver cancer.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Primary Liver Cancer: Patients that have liver masses suspicious for primary liver cancer.

SUMMARY:
To collect tumor tissue from patients with liver masses suspicious for primary liver cancer. The research biopsy will be used to identify biomarkers in future studies.

DETAILED DESCRIPTION:
In this study patients are referred to the Department of Radiology for an image-guided (either CT or ultrasound) core needle biopsy of a liver mass suspicious for primary liver cancer as a part their clinical care. A written informed consent will be obtained for the clinical biopsy per standard protocol. Additional core biopsy of the liver mass will be performed for research purposes at the time of the clinical care biopsy. The additional research biopsy is not mandatory and is subject to a separate written informed consent, which will be obtained prior to the clinical biopsy.

ELIGIBILITY:
Inclusion Criteria:

1. Liver mass suspicious for primary liver cancer with a diagnostic liver biopsy planned as a part of clinical care
2. Age ≥ 18 years.
3. ECOG performance status 0-2
4. Adequate organ and marrow function as defined below:

   INR ≤ 1.5 platelets ≥ 70,000/mcl
5. Ability to understand and the willingness to sign a written informed consent
6. Target liver mass not subcapsular in nature as determined by the participating biopsy team
7. Child Pugh Turcotte score A or B

Exclusion Criteria:

1. Previous treatment for HCC
2. Any contraindication for clinical-care liver biopsy, including anti-coagulation therapy that cannot be discontinued prior to biopsy or large volume ascites

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 500 patients with a liver mass suspicious for HCC
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-10; Primary Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Biopsy of Liver Masses | 5 years
  To obtain tissue from biopsy of liver masses suspicious for primary liver cancer for use in future biomarker studies.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Yopp, MD, Principal Investigator — University of Texas Southwestern Medical Center